CLINICAL TRIAL: NCT03241420
Title: Utility of Lung Clearance Index Score As a Noninvasive Marker of Small Airways Disease
Status: Active, not recruiting | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Cecile Rose Professor of Medicine, PI, National Jewish Health
Other Study IDs: HS-2985
Record Dates: First submitted 2017-07-24; First posted 2017-08-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Chronic Lung Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic Lung conditions: Study participation will consist of one visit: Informed consent, complete both Lung Clearance Index (LCI) testing and spirometry.
  Interventions: Device: lung clearance index (LCI)
- Healthy control group: Study participation will consist of one visit: Informed consent, brief questionnaire, LCI testing and spirometry.
  Interventions: Device: lung clearance index (LCI)

INTERVENTIONS:
Device: lung clearance index (LCI) — Determine the utility and sensitivity of the lung clearance index (LCI) technique as a marker of lung injury/small airways disease in adults with chronic lung conditions compared to health adults, adjusting for age, sex, and smoking status.

SUMMARY:
To determine the utility and sensitivity of the lung clearance index (LCI) technique as a marker of small airways disease in adults with chronic lung conditions compared to healthy adults, adjusting for age, sex and smoking status.

DETAILED DESCRIPTION:
Target Population and Enrollment. The study will recruit and consent 300 patients from our Occupational Medicine and Interstitial Lung/Rheumatology Clinics at National Jewish Health who have been referred for evaluation of chronic lung conditions. The healthy control group will comprise 300 volunteers who are at least 18 years of age, have no history of pre-existing lung disease, and report no respiratory illness in the four weeks preceding enrollment. Inclusion criteria for the group with chronic lung disease will include physician diagnosis of a chronic lung condition (e.g. bronchiolitis, pulmonary fibrosis, asthma, coal mine dust lung disease, asbestosis), and age ≥18 years. Exclusion criteria will include recent myocardial infarction, stroke, eye surgery, chest/abdominal surgery (within past month), known thoracic, aortic, or cerebral aneurysm, or uncontrolled hypertension. Study participation will consist of one visit that will last between 90-120 minutes. The chronic lung disease group will fill out the informed consent and complete both LCI testing and spirometry. The healthy control group will complete informed consent, a brief questionnaire, LCI testing, and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of a chronic lung condition (e.g. bronchiolitis, pulmonary fibrosis, asthma, coal mine dust lung disease, asbestosis), and age ≥18 years.

The healthy control group will comprise 300 volunteers who are at least 18 years of age, have no history of pre-existing lung disease, and report no respiratory illness in the four weeks preceding enrollment

Exclusion Criteria:

* Exclusion criteria will include recent myocardial infarction, stroke, eye surgery, chest/abdominal surgery (within past month), known thoracic, aortic, or cerebral aneurysm, or uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Symptomatic military deployers with deployment-related lung disease seen at National Jewish Health and healthy controls subjects.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lung Clearance Index (LCI) technique can be used as a marker of small airways disease in adults with chronic lung conditions | Up to 12 months
  Average of three acceptable trials.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Zell-Baran LM, Krefft SD, Moore CM, Wolff J, Meehan R, Rose CS. Multiple breath washout: A noninvasive tool for identifying lung disease in symptomatic military deployers. Respir Med. 2021 Jan;176:106281. doi: 10.1016/j.rmed.2020.106281. Epub 2020 Dec 5. PMID 33340829
- [Background] Zell-Baran LM, Krefft SD, Moore CM, Wolff J, Meehan R, Rose CS. Multiple breath washout test data for healthy controls. Data Brief. 2020 Dec 10;34:106641. doi: 10.1016/j.dib.2020.106641. eCollection 2021 Feb. PMID 33365370